CLINICAL TRIAL: NCT00258778
Title: A Phase I, Non-Randomized, Open Label, Single Dose-Escalation Safety Study of Recombinant Human Glucocerebrosidase (prGCD) in Healthy Volunteers
Brief Title: Phase I Single Dose-Escalation Safety Study of Human Glucocerebrosidase (prGCD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Protalix (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-01-2005
Record Dates: First submitted 2005-11-23; First posted 2005-11-28 (Estimated); Last update posted 2006-12-05 (Estimated); Status verified 2006-12

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease | interventions — taliglucerase alfa

INTERVENTIONS:
Drug: Human Glucocerebrosidase (prGCD)

SUMMARY:
Gaucher disease, the most prevalent lysosomal storage disorder, is caused by mutations in the human glucocerebrosidase gene (GCD)leading to reduced activity of the lysosomal enzyme glucocerebrosidase and thereby to the accumulation of substrate glucocerebroside (GlcCer)in the cells of the monocyte-macrophage system.

This is the first trial to utilize a recombinant active form of lysosomal enzyme, glucocerebrosidase, (human prGCD)which is expressed and purified in a bioreactor system from transformed carrot plant root cell line.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female between 18 and 45 years of age.
2. Female subjects must agree to use a medically acceptable method of contraception at all times during the study and must have a negative serum pregnancy test at baseline and during the study period.
3. Females of child-bearing potential must be non-pregnant and not lactating and using adequate birth control such as oral contraceptives.
4. Negative laboratory tests for HIV, HBsAg or HCV.
5. Naive to any previous recombinant protein therapy.
6. Provide written informed consent.
7. Have the ability to understand the requirements of the study and to comply with the study protocol and dosing regimen.

Exclusion Criteria:

1. Have clinical evidence of any active significant disease that could potentially compromise the ability of the investigator to evaluate or interpret the effects of the study treatment on safety assessment and thus increase the risk to the subject to unacceptable levels.
2. Are pregnant or nursing.
3. Presence of any acute or chronic diseases.
4. Have a history of any allergies.
5. Have been exposed to long-term steroid treatment.
6. Had a minor operation in the last 6 months.
7. Have ever been exposed to any previous recombinant protein therapy.
8. Have received immuno-suppressive treatment.
9. Have a positive HIV, HBsAG and HCV laboratory result.
10. Use any medication other than vitamins or oral contraceptives (for female).
11. Have participated in another clinical trial during the previous 3 months
12. Have history of alcohol or drug abuse.
13. Are considered by the Investigator to be unsuitable candidate for this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6
Dates: Start 2005-11; Study Completion 2006-01

PRIMARY OUTCOMES:
Safety as measured by:
adverse events
change in vital signs
physical examination
laboratory test results

SECONDARY OUTCOMES:
Pharmacokinetic parameters
Immunological profile including: IgE, anti human prGCD antibodies, eosinophils and proteinuria

CONTACTS AND LOCATIONS:
Overall Officials: Eithan Galun, MD, Principal Investigator — Protalix Ltd.

REFERENCES:
- [Derived] Aviezer D, Brill-Almon E, Shaaltiel Y, Hashmueli S, Bartfeld D, Mizrachi S, Liberman Y, Freeman A, Zimran A, Galun E. A plant-derived recombinant human glucocerebrosidase enzyme--a preclinical and phase I investigation. PLoS One. 2009;4(3):e4792. doi: 10.1371/journal.pone.0004792. Epub 2009 Mar 11. PMID 19277123